CLINICAL TRIAL: NCT02089503
Title: Monocentric Retrospective Observational Study Describing the Visual Acuity of Patients With Exudative Age Related Macular Degeneration and Treated by Lucentis® Under Real Conditions of Care.
Brief Title: Monocentric Retrospective Observational Study on Patients With Macular Degeneration
Acronym: ELOUAN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, QUEGUINER, MD, Ophtalmologist, Hospital St. Joseph, Marseille, France
Other Study IDs: ELOUAN HSJ 2014
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Exudative Age-Related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- induction phase + intravitreal inj.: Group of patients who received Lucentis ® with induction phase
  Interventions: Other: intravitreal injections of Lucentis
- intravitreal inj. without induction: Group of patients who received Lucentis ® without induction phase
  Interventions: Other: intravitreal injections of Lucentis
- intravitreal inj. + monthly follow-up: group of patients who were monthly monitored (+/- 1 week)
  Interventions: Other: intravitreal injections of Lucentis
- intravitreal inj. + follow-up :> 1 month: group of patients with Follow up visits intervals> 1 month (+/- 1 week)
  Interventions: Other: intravitreal injections of Lucentis
- intravitreal inj +induction+ month. FU: Group of patients who received Lucentis with induction phase and who were monthly monitored (+/- 1 week)
  Interventions: Other: intravitreal injections of Lucentis
- date Lucentis® 1st intravitreal Inj.: Group of patients selected in accordance with the date of Lucentis® treatment start.
  Interventions: Other: intravitreal injections of Lucentis

INTERVENTIONS:
Other: intravitreal injections of Lucentis — intravitreal injections FOR ALL PATIENTS of Lucentis as required in the normal condition of use

SUMMARY:
Main Objective: The main objective of this retrospective observational study was to describe the evolution of visual acuity measured on ETDRS (Early Treatment Diabetic Retinopathy Study) scale, for patients with exudative Age-Related Macular Degeneration (ARMD), treated with Lucentis, under real conditions of care, in terms of mean change of the Best Corrected Visual Acuity (BCVA), measured at 24 months (± 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients with exudative-subfove ARMD, regardless the neovessel type or the initial visual acuity; 2 - Patients treated in the department with intra vitreous injection of Lucentis ® during the study period (08/2011 and 02/2013); 3 - If both eyes are eligible, both will be analyzed;

Exclusion Criteria:

1. - Patients who received, for the studied eye, a treatment with a Vascular endothelial growth factor (VEGF) other than Lucentis ® in the three months preceding the start of the study. For those who received combination therapy, the nature of the treatment will be specified and taken into account in the subgroups for statistical analyzes;
2. - Patients with high myopia or neovessel not related to exudative-ARMD;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with exudative Age-Related Macular Degeneration (ARMD), treated with Lucentis, under real conditions of care
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA), measured at 24 months (± 4 weeks). | measured at 24 months (± 4 weeks)

SECONDARY OUTCOMES:
the mean change of the BCVA throughout the 24 months of follow-up (FU), | 24 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maud RIGHINI, MD, Study Chair — HSJ
Locations (1):
- Hopital Saint Joseph, Marseille, France